CLINICAL TRIAL: NCT03851263
Title: Multi-slice CT Scan Assessment of the Impact of PCSK9 Inhibition With Evolocumab on Coronary Perfusion in Patients With Reduced Coronary Fractional Flow Reserve (FFR).
Brief Title: Multislice Computed Tomography Assessment of PCSK9 Inhibition on Coronary Perfusion
Acronym: MARKOV
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Admisnitrative issues
Sponsor: ECRI bv (Industry)
Collaborators: Amgen (Industry); GE Healthcare (Industry); HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECRI-11
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evolocumab (Experimental): All subjects are treated with evolocumab 140mg every 2 weeks (q2w) starting on day 1 and ending on day 1071 (week 153).
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Subcutaneous injection, using a pre-filled auto-injector pen. Each pen contains 1.0 ml fluid (containing 140 mg evolocumab) which is injected in the abdomen, thigh or outer area of upper arm every 2 weeks (q2w).

SUMMARY:
The MARKOV study is an investigator-sponsored single arm, prospective study to assess the effect of evolocumab on the improvement in coronary flow (FFRCT) after 18 and 36 months of treatment in patients with coronary atherosclerosis.

DETAILED DESCRIPTION:
The MARKOV study is an investigator-initiated, open-label, single arm, international, multicenter, prospective study to assess the effect of evolocumab on the improvement in coronary flow (FFRCT) after 18 and 36 months of treatment in patients with coronary atherosclerosis. The study will be conducted in 5 sites in 3 different countries in Europe. Patients will receive evolocumab for approximately 3 year. The expected duration of the entire study from First Subject First Visit to Last Subject Last Follow-up is 46 months (3 year and 10 months).

ELIGIBILITY:
Inclusion Criteria:

1. At least 2 coronary vessels suitable for CCTA; vessels fulfilling all requirements below: a. patent main branch b. no previous stent placement
2. At least two of the evaluable vessels with subclinical coronary artery disease as defined non-invasively by CCTA with encroachment of the vessel and either: a. Lesion with visual diameter stenosis (DS) < 50% or, b. Lesion with visual DS ≥ 50% and FFRCT > 0.80;
3. No planned coronary revascularization (during the course of the study) at the time of enrollment;
4. Most recent, taken within 30 days prior to informed consent form (ICF) signature, fasting LDL-C ≥ 80 mg/dL (≥ 2.07 mmol/L) and on stable statin therapy for at least 30 days at the time of blood sampling, or statin-intolerant or for whom a statin is contraindicated.
5. Subject signed informed consent form

Exclusion Criteria:

1. History of coronary artery bypass surgery, heart transplantation, surgical or percutaneous valve repair and/or replacement
2. New York Heart Association (NYHA) class III or IV heart failure
3. Last known left ventricular ejection fraction <30%
4. Active liver disease or hepatic dysfunction, either known or defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 times the upper limit of normal (ULN)
5. Severe renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2
6. Active malignancy except for adequately treated non-melanoma skin cancer or other non-invasive or in situ neoplasm (e.g. successfully treated cervical cancer in situ or non-active prostate cancer) Imaging CCTA-related
7. Absence of baseline CCTA obtained in the context of standard clinical care
8. Baseline CCTA not meeting Core Lab quality standards
9. Any contraindication for repeat CCTA such as known anaphylactic allergy to iodinated contrast

   Concomitant and study medication
10. Any prior or current use of PCSK9 inhibition treatment or any other experimental lipid-related drug Other exclusion criteria
11. LDL or plasma apheresis within 12 months of screening
12. Subject < 18 years of age
13. Legally incompetent to provide written informed consent;
14. Known pregnancy or breast-feeding at time of screening
15. Female subject of childbearing potential, i.e. who are not surgically sterile or post-menopausal (defined as no menses for 2 years without an alternative cause)
16. Male subject with female partner of childbearing potential who is not using highly effective birth control
17. Currently participating in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2021-08-27 (Estimated); Study Completion 2023-02-24 (Estimated)

PRIMARY OUTCOMES:
Mean change in normalized area under the curve of fractional flow reserve derived from coronary computed tomography(CCTA) (FFRCT) at 18 months from baseline | 18 months of treatment

SECONDARY OUTCOMES:
Mean change in normalized area under the curve of fractional flow reserve derived from coronary computed tomography (FFRCT) at 36 months from baseline. | 36 months of treatment
Percent change of total atheroma burden (TAB) and changes in plaque composition at 18 and 36 months measured by Hounsfield unit of plaque with positive remodeling (>1.10) assessed by coronary computed tomography. | 18 and 36 months of treatment
Change and percent change after 18 and 36 months from baseline of total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL), lipoprotein (a), triglycerides, apolipoprotein A1 and B. | 18 and 36 months of treatment
Number of treatment emergent adverse events (TEAEs) and adverse events (AEs) of special interest (i.e. acute kidney injury, pregnancy and lactation) | 36 months of treatment
Incidence of all-cause death and the composite of Cardiovascular death, myocardial infarction, stroke, or coronary revascularization. The composite of Cardiovascular death, Myocardial infarction, or stroke | 36 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, Prof. dr., Study Chair — NHLI Imperial College, London

IPD SHARING:
Plan to Share IPD: Undecided